CLINICAL TRIAL: NCT00669916
Title: Phase 2a Single-Dose, Randomized, Double Blind, Multi-Center, Parallel-Group, Placebo-Controlled Proof of Concept Study to Assess the Efficacy, Safety, Tolerability, and Population Pharmacokinetics of AIN457 in Patients With Stable Plaque-type Psoriasis
Brief Title: A Study Comparing AIN457 to Placebo in Subjects With a Diagnosis of Moderate to Severe Stable Plaque Psoriasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CAIN457A2102
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Plaque Psoriasis
Keywords: Plaque psoriasis
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIN457 (Experimental): AIN457A 3mg/kg was administered intravenously as a single dose.
  Interventions: Biological: AIN457
- Placebo (Placebo Comparator): Placebo was administered intravenously as a single dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AIN457 — single infusion of 3 mg/kg
  Arms: AIN457
Drug: Placebo — single infusion of placebo
  Arms: Placebo

SUMMARY:
This is a two-arm, parallel group, double-blind, placebo-controlled proof-of-concept study comparing 3 mg/kg of AIN457 to placebo. Subjects with a diagnosis of moderate to severe stable plaque psoriasis will be randomized to receive either AIN457 or placebo. AIN457 or placebo will be administered by single infusion at baseline and subjects will be observed for up to 26 weeks following the infusion.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged 18-69 at time of consent.
* Post menopausal or surgically sterile female patients are allowed. Male patients must be willing to use contraception method at least for 3 months following the completion of the study. Women of child-bearing potential will not be allowed to participate.
* Diagnosis of plaque psoriasis for at least 6 months prior to screening. The patients must meet both of the following criterion:

  1. Coverage of the body surface area (BSA) of 10% or more with plaques
  2. A score of 3 or more on the IGA scale
* Stable plaque psoriasis at screening and randomization.
* PASI score of 12 or greater at randomization.
* Able to communicate well with the investigator, and to understand and comply with the requirements of the study. Understand and sign the written informed consent.
* Patients must have normal laboratory values for screening laboratory test results of hematological (hemoglobin, WBCs, neutrophils, platelets) and renal (serum creatinine) assessments. For the transaminases, aspartate aminotransferase and alanine aminotransferase, levels 1.5 times the upper limit of normal will be accepted. For the additional hepatic laboratory results (alkaline phosphatase, gamma-glutamyltransferase, bilirubin), patients must have non-clinically significant values.

Exclusion Criteria:

* Currently have any of the nonplaque forms of psoriasis: erythrodermic, guttate, or pustular.
* Currently have drug-induced psoriasis (new onset or exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium).
* Men who are planning to initiate a pregnancy while enrolled in the study or for 3 months following completion of the study.
* Women of child-bearing potential are not allowed in the study.
* Used any investigational drug within the previous 4 weeks.
* Recent previous treatment with anti-TNF-α therapy (or other biological therapy), immunosuppressive agents such as cyclosporine, mycophenolate, pimecrolimus, or tacrolimus. The following washout period will be required for such patients to be eligible to participate in the trial.

  1. 2 months washout prior to screening for etanercept, adalimumab, or infliximab.
  2. 1 month washout prior to screening for cyclosporine, mycophenolate, tacrolimus, and any systemic immunosuppressants including, but not limited to, methotrexate, azathioprine, 6-thioguanine, mercaptopurine, and hydroxyurea

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

REFERENCES:
- [Derived] Hueber W, Patel DD, Dryja T, Wright AM, Koroleva I, Bruin G, Antoni C, Draelos Z, Gold MH; Psoriasis Study Group; Durez P, Tak PP, Gomez-Reino JJ; Rheumatoid Arthritis Study Group; Foster CS, Kim RY, Samson CM, Falk NS, Chu DS, Callanan D, Nguyen QD; Uveitis Study Group; Rose K, Haider A, Di Padova F. Effects of AIN457, a fully human antibody to interleukin-17A, on psoriasis, rheumatoid arthritis, and uveitis. Sci Transl Med. 2010 Oct 6;2(52):52ra72. doi: 10.1126/scitranslmed.3001107. PMID 20926833

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AIN457 | Placebo
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.7 (8.73) | 50.9 (12.04) | 50.8 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Mean Score
Description: The PASI assessed the extent of psoriasis on four body surface areas (head, trunk and upper limbs) and the degree of plaque erythema, scaling and thickness. The PASI score accounted for the extent of body surface area affected by the erythema, scaling and thickness and the severity of these measures. The score ranged from 0 (no disease) to 72 (maximal disease) where a reduction in PASI score from baseline indicates improvement. The percentage change was calculated by subtracting the week 4 values from the baseline values.The percentage change was calculated for each entire treatment group (not for each participant). A positive percentage change from baseline indicates improvement.
Time Frame: Baseline, Week 4
Population: All participants
Measure: Number; unit: Percentage change in PASI mean score
Arm/Group | AIN457 | Placebo
Number analyzed (Participants) | 18 | 18
Percentage change in PASI mean score | 58 | 4

2. Secondary Outcome: Pharmacokinetics of AIN457: Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: Blood was drawn for PK analyses at baseline (prior to dosing), end of infusion, 1 hr and 2 hr after infusion, and during office visits in Weeks 1, 2, 3, 4, 5, 6, 8, 12, 16, 20 and 26. The PK samples may have been taken at any time during each office visit, following the day of study drug infusion. This outcome measure shows the mean of all values resulting from each time point outlined above.
Time Frame: Day 182
Population: The population included all AIN457 treatment group participants except for two participants who had a nontypical PK profile for Tmax, Cmax, CI and Vz.
Measure: Median (Full Range); unit: days
Arm/Group | AIN457
Number analyzed (Participants) | 16
days | 0.11 [0.08 to 0.17]

3. Secondary Outcome: Pharmacokinetics of AIN457: Observed Maximum Serum Concentration Following Drug Administration (Cmax)
Description: as for outcome 2
Time Frame: Day 182
Population: The population included all AIN457A treatment group participants except for two participants who had a nontypical PK profile for Tmax, Cmax, CI and Vz.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | AIN457
Number analyzed (Participants) | 16
ug/mL | 74.5 (13.1)

4. Secondary Outcome: Pharmacokinetics of AIN457: Area Under the Serum Concentration-time Cure From Time Zero to the Time of Last Quantifiable Concentration (AUClast), Area Under the Serum Concentration-time Curve From Time Zero to (AUCinf)
Description: as for outcome 2
Time Frame: Day 182
Population: All AIN457A treatment group participants
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | AIN457
Number analyzed (Participants) | 18
day*ug/mL
  AUClast | 1532 (343)
  AUCinf | 1629 (361)

5. Secondary Outcome: Pharmacokinetics of AIN457: Volume of Distribution During the Terminal Phase Following Intravenous Elimination (Vz)
Description: as for outcome 2
Time Frame: Day 182
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Liters
Arm/Group | AIN457
Number analyzed (Participants) | 16
Liters | 7.31 (1.72)

6. Secondary Outcome: Pharmacokinetics of AIN457: Systemic Clearance From Serum Following Intravenous Administration (CL)
Description: as for outcome 2
Time Frame: Day 182
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liters/day
Arm/Group | AIN457
Number analyzed (Participants) | 16
Liters/day | 0.18 (0.05)

7. Primary Outcome: Percentage of Participants With Change From Baseline in Investigators Global Assessment (IGA) Score
Description: The IGA is an instrument which captured and categorized the global assessment of all clinical signs and symptoms of disease. The investigator used all available information for the assessment, including subjective information from the participant and (where available) photographs taken at baseline. The IGA categories were clear, almost clear, mild disease, moderate disease, severe disease and very severe disease. This outcome measure shows the percentage of patients who experienced a category change from baseline. Category changes of 1, 2 or 3 indicate improvement.
Time Frame: Baseline, Week 4
Population: All participants
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 | Placebo
Number analyzed (Participants) | 18 | 18
Percentage of participants
  Change in IGA score = -1 | 5.6 | 11.1
  Change in IGA score = 0 | 11.1 | 77.8
  Change in IGA score = 1 | 33.3 | 11.1
  Change in IGA score = 2 | 44.4 | 0
  Change in IGA score = 3 | 5.6 | 0

8. Secondary Outcome: Pharmacokinetics of AIN457: Terminal Elimination Half-life (T1/2)
Description: as for outcome 2
Time Frame: Day 182
Population: All AIN457A treatment group participants
Measure: Mean (Standard Deviation); unit: day
Arm/Group | AIN457
Number analyzed (Participants) | 18
day | 29.2 (6.4)

ADVERSE EVENTS:
Groups:
- AIN457A: AIN457A 3mg/kg was administered intravenously as a single dose.
Arm/Group | AIN457A | Placebo
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18
Other Adverse Events (participants affected / at risk) | 9/18 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457A (N=18) | Placebo (N=18)
Cardiac failure congestive (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457A (N=18) | Placebo (N=18)
Corneal degeneration (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Injection site infection (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 2 | 1
Blood ketone body increased (Investigations) | 1 | 0
Blood triglycerides increased (Investigations) | 2 | 2
Glucose urine present (Investigations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Protein urine present (Investigations) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin maceration (Skin and subcutaneous tissue disorders) | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.